CLINICAL TRIAL: NCT04412447
Title: Training of Persons With Complete Spinal Cord Injury for Pedaling on a Tricycle, Induced by Electrical Stimulation of the Paralysed Muscles: a Case Series
Brief Title: Training for Persons With Complete SCI for FES Cycling: a Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre de Rééducation et Réadaptation Fonctionnelle La Châtaigneraie (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other); Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-A00808-49
Record Dates: First submitted 2020-05-11; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Training of paralysed musculature of the lower limb by using electrical stimulation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Experimental): Phase V1: 1 month of home-based FES-training using isometric contractions of quadriceps and hamstring muscles (3 times a week).
  Phase V2: 2 months of home-based FES-training on an ergo-cycle with arm support (3 times a week)
  Phase V3: 1 month of home-based FES-training on an ergo-cycle with arm support (1-2 times a week) and FES-cycling training overground on a tricycle (1-2 times a week) in the clinical setting.
  Optional (only for selected pilot):
  Phase V4: 2-4 months of home-based FES-training on an ergo-cycle with arm support (1-2 times a week) and FES-cycling training overground on a tricycle (1-2 times a week) in the clinical setting. This phase is focussing on optimizing the performance of the pilot and improving the mechanical efficiency of the tricycle.
  Phase V5: Participation on Cybathlon 2020
  Interventions: Device: Functional Electrical Stimulation

INTERVENTIONS:
Device: Functional Electrical Stimulation — Electrical stimulation of motor-nerves innervating the musculature of the lower limb.

SUMMARY:
The main objective of this study is to validate the effectivity of a simple home-based training for cycling with functional electrical stimulation (FES). The training is designed to progressively increase strength and endurance of the paralysed muscles of a person with complete spinal cord injury. After a limited period of only several months, performance will be assessed during FES-assisted cycling on a recumbent tricycle over flat ground. The outcomes of this study should provide evidence for the effectivity of FES-cycling as potential rehabilitation method.

DETAILED DESCRIPTION:
People with spinal cord injuries suffer from numerous comorbidities, linked in particular to immobility and sedentariness. Studies have shown the benefits of training and reconditioning to adapted effort in spinal cord injured people. Among other innovative techniques, functional electrical stimulation (FES) is aimed primarily at mobilizing as many muscles as possible. Concerning electro-stimulated pedaling on a tricycle, it would allow individuals with paraplegia or tetraplegia to practise physical activity in perspective of experiencing pleasure during training.

In 2016, our team carried out a pilot study aiming at using a recumbent tricylce powered by the lower limbs of a person with complete paraplegia under electrostimulation. The participant was trained for 12 months, whit the objective to participate at an international competition (Cybathlon 2016). This first study has opened up prospects and identified avenues for improvement.

The main objective of this study is to significantly improve, over a limited period of time, the pedalling performance on a tricycle by using electrical stimulation of the sub-lesional muscles of people with spinal cord injuries. Secondary focusses will be: physical and psychological tolerance to training; influence on pain, cardio-respiratory functions, body composition regarding muscle trophicity and bone metabolism; psycho-social impact; impact of modification of stimulation parameters (frequency, phase width, intensity, waveform, contact location) in performance optimization and delay of muscle fatigue; performance impact of mechanical modifications performed on the tricycle.

This is a prospective case study: patients suffering from a complete traumatic injury and followed at the Centre de Rééducation et de Réadaptation Fonctionnelle (CRRF) La Châtaigneraie (Menucourt) will be recruited by the investigating physician during a consultation for a period of approximately 6 months. The centre specialised in the management of acute and chronic neurological lesions. The eligibility criteria are predefined to ensure the participants safety. After verification of the criteria and before the start of the programme, an exercise test (monitoring of the evolution of VO2max) will be carried out in the Sports Medicine department of the CHI of Saint-Germain-en-Laye. The first phase (V1) consists of a one-month home-based isometric muscle training programme by electrostimulation followed by a two-month programme (phase V2) of home-based muscle training by electrostimulation on an ergocycle including one training per week at the CRRF. The home ergocycle electro-stimulation muscle training, will be continued once or twice a week and complemented in the third phase (V3) by training at the CRRF on a tricycle for one month. Only the patient selected to participate in the Cybathlon 2020 will continue with the final phase (V4), which includes, over a period of 2 to 4 months, muscle training by electrostimulation on an ergocycle at home, electrostimulation sessions on a tricycle up to 3 times a week at the CRRF. In this phase, the optimization of the stimulation and electrical patterns and the mechanics of the tricycle will take place in order to maximize the pilots overall performance. Finally, the pilot will take part in the tricycle FES-Cycling race at the Cybathlon 2020 in Zurich, i.e. an international competition and technological challenge, requiring to master 1200 metres in a maximum time of 8 minutes. The different training programs are based on sport-scientific principles and a physiotherapist will follow up on the home sessions. The collaborating teams (engineers and researchers from INRIA, the French National Institute for Research in Computer Science and Control) will measure performance in a bimonthly frequency.

This research should demonstrate that the safety, acceptability, satisfaction, self-esteem and quality of life induced by the practice of FES-assisted pedalling, opens a new way of training in rehabilitation centres and at home with the perspective of improving certain physiological functions in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent
* complete spinal cord injury AIS A or B
* neurological level of lesion C6 - T12
* post-lesion duration > 12 moths
* paralysed muscles stimulable
* joints of lower limb freely moveable
* stable medical condition (absence of infectious respiratory or urinary event of cutaneous pathology confining the patient to bed and warranting treatment).

Exclusion Criteria:

* Not affiliated to a social security scheme, beneficiary or not such a plan
* Refusal to participate in the study (withdraw from study possible at any time)
* Inability to give consent
* body mass index higher or equal to 30
* flaccid paralysis (denervation)
* Inability to give consent
* neurogenic para-osteoarthropathy
* active thrombophlebitis
* muscular disease
* cardiovascular disease including coronary antecedent
* bone mineral density T-score below -2.5
* treatment with a drug known to have an effect on bone (< 3 months)
* Aids in the lower limbs
* Epilepsy
* Orthostatic hypotension
* Fractures of the lower limbs older (< 12 months)
* Pacemakers or other implants contraindicating the use of FES
* Pregnancy (women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in Maximum Cycling-Distance in [m] | Change between 4 months of training (end of V3) and 6 months of training (end of V4)
  Change in maximum distance cycled on flat ground on a tricycle
Change in Maximum Cycling-Speed in [km/h] | Change between 4 months of training (end of V3) and 6 months of training (end of V4)
  Change in maximum speed during cycling over flat ground on a tricycle
Change in Average Cycling-Speed in [km/h] | Change between 4 months of training (end of V3) and 6 months of training (end of V4)
  Change in average speed during cycling over flat ground on a tricycle
Change in Maximum Cycling-duration in [hh:mm:ss] | Change between 4 months of training (end of V3) and 6 months of training (end of V4)
  Change in maximum duration during cycling over flat ground on a tricycle
Change in Maximum Pedaling-Cadence in [RPM] | Change between 4 months of training (end of V3) and 6 months of training (end of V4)
  Change in maximum pedaling-cadence during cycling over flat ground on a tricycle
Change in Average Pedaling-Cadence in [RPM] | Change between 4 months of training (end of V3) and 6 months of training (end of V4)
  Change in average pedaling-cadence during cycling over flat ground on a tricycle
Ability to cycle 1200m in less than 8min | After 6 months of training (end of V4)
  Qualification criterion Cybathlon 2020. It will be assessed it the pilot is able to cycle 1200m in less than 8min over flat ground on a tricycle.

SECONDARY OUTCOMES:
Change of blood pressure during training | through study completion (up to one year), an average throughout the study-duration
  Blood pressure will be assessed before and after every training session. Mean change in blood pressure will be calculated along all training-sessions.
Change of heart rate during training | through study completion (up to one year), an average throughout the study-duration
  Heart rate will be assessed before and after every training session. Mean change in heart-rate will be calculated along all training-sessions.
Maximum heart rate during training | through study completion (up to one year), an average throughout the study-duration
  Maximum heart rate will be assessed during every training session. Mean and SD of the maximum heart-rate will be calculated along all training-sessions.
Average heart rate during training | through study completion (up to one year), an average throughout the study-duration
  Average heart rate will be assessed during every training session. Mean and SD of the average heart-rate will be calculated along all training-sessions.
Cutaneous status | through study completion (up to one year)
  Evaluation for absence of: skin lesions, pressure points, pressure ulcers, phlebitis, edema
Musculo-skeletal pain or inflammation | through study completion (up to one year)
  Evaluation for absence of: muscular pain, osteo-articular pain or inflammation
Psychological: Satisfaction | through study completion (up to one year), an average throughout the study-duration
  Evaluation of satisfaction [linear scale: 1 - 10; 1 = lowest satisfaction; 10 = highest satisfaction] will be assessed after every training session. Mean and SD of the satisfaction will be calculated along all training-sessions.
Psychological: Acceptability | through study completion (up to one year), every 30 days
  Change in acceptability [questionnaire].
General Fatigue | through study completion (up to one year), an average throughout the study-duration
  Assessment of change in general fatigue via [Borg scale; Range: 6-20; 6 = No exertion, sitting and resting; 20 = Maximal exertion] will be assessed before and after every training session. Mean and SD of the change in fatigue will be calculated along all training-sessions.
Psycho-Social: Self-Esteem | through study completion (up to one year), every 15 days
  Change in self-esteem via [Rosenberg Scale; Range: 10 - 40; 10 = lowest Self-Esteem; 40= Highest Self-Esteem].
Psycho-Social: Quality of Life | through study completion (up to one year), every 30 days
  Change in quality-of-life via [questionnaire SF-36].
Cardio-Respiratory Fitness: Maximal Heartrate | Change between timepoint before first training, after 4 months of training (end of V3) and after 6 months of training (end of V4)
  Change of maximal heartrate via electrocardiogram
Cardio-Respiratory Fitness: VO2max | Change between timepoint before first training, after 4 months of training (end of V3) and after 6 months of training (end of V4)
  Change of VO2max
Musculo-skeletal changes: Thigh perimeter | Change between timepoint before first training and after end of study (end of V5, ~ 7 months)
  Assessment of thigh perimeter [cm]. Measurement is taken 10cm and 20cm proximal to the proximal edge of the patella.
Musculo-skeletal changes: Bone mineral density | Change between timepoint before first training and after end of study (end of V5, ~ 7 months)
  Bone mineral density via [DEXA]
Musculo-skeletal changes: Body composition | Change between timepoint before first training and after end of study (end of V5, ~ 7 months)
  Body composition via [DEXA].
Occurrence of spasms: before training | through study completion (up to one year), an average throughout the study-duration
  Spasmic occurance will be assessed via [PENN Scale; Range: 0-4; 0 = No spasm; 4 = Spasms occuring more than 10 times per hour] before every training session. Mean and SD of the spasmic occurence will be calculated along all training-sessions.
Occurrence of spasms : after training | through study completion (up to one year), an average throughout the study-duration
  Spasmic occurance will be assessed via [PENN Scale; Range: 0-4; 0 = No spasm; 4 = Spasms occuring more than 10 times per hour] after every training session. Mean and SD of the spasmic occurence will be calculated along all training-sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Rééducation et de Réadaptation Fonctionnelle La Châtaigneraie, Menucourt, France

REFERENCES:
- [Derived] Fattal C, Schmoll M, Le Guillou R, Raoult B, Frey A, Carlier R, Azevedo-Coste C. Benefits of 1-Yr Home Training With Functional Electrical Stimulation Cycling in Paraplegia During COVID-19 Crisis. Am J Phys Med Rehabil. 2021 Dec 1;100(12):1148-1151. doi: 10.1097/PHM.0000000000001898. PMID 34596097